CLINICAL TRIAL: NCT06509009
Title: Nimotuzumab Combined With Toripalimab/Gemcitabine/Cisplatin as First-line Therapy in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma: a Prospective, Single-arm, Phase II Clinical Study
Brief Title: Nimotuzumab Combined With TGP as First-line Therapy in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TINPC-001
Record Dates: First submitted 2024-05-23; First posted 2024-07-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage
Keywords: nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab combine with TGP (Experimental): Base on TGP(Toripalimab, Gemcitabine, and Cisplatin) regimen, the patients will receive Nimotuzamab treatment.
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — nimotuzumab, toripalimab, gemcitabine, cisplatin
  Other Names: no other invention names

SUMMARY:
The goal of this study is to learn the efficacy and safety of nimotuzumab combined with toripalimab and gemcitabine/cisplatin regimen treatment recurrent/distant-metastasis nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The study is to investigate the efficacy and safety of combining nimotuzumab and toripalimab with the GP regimen for first line recurrent/distant metastasis nasopharyngeal carcinoma.

This clinical trial adopts a single-center, prospective, single-arm phase II trial design. Each treatment cycle will be three weeks long, the chemotherapy regimen contains no more than 6 circles, nimotuzumab and toripalimab were used until progression.

After screening, eligible patients will be enrolled in the study. Patients will receive up to 6 cycles of nimotuzumab and toripalimab, gemcitabine, cisplatin therapy. Patients will undergo regular follow-up visits, and researchers will collect data on efficacy and safety. Short-term outcomes will be assessed according to the RECIST 1.1 criteria/irRECIST, and adverse events will be evaluated using the CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent form.

Age between 18 and 75 years, inclusive, without gender restriction.

Histologically confirmed diagnosis of recurrent/distant metastasis nasopharyngeal carcinoma, first line patients and unsuitable for local operation treatment.

EGFR expression positive.

Presence of at least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and patients who have not undergone definitive treatment.

ECOG Performance Status (PS) score of 0 or 2.

Expected survival duration of at least 3 months.

White blood cell count ≥ 3 × 10^9/L; absolute neutrophil count ≥ 1.5 × 10^9/L; platelet count ≥ 100 × 10^9/L; hemoglobin level ≥ 90 g/L.

Serum creatinine level ≤ 1.2 mmol/L or creatinine clearance ≥ 60 ml/min.

Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (in case of liver metastasis, ≤ 3.0 × ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (in case of liver metastasis, ≤ 5.0 × ULN).

Female patients must have a negative urine pregnancy test prior to study enrollment (this criterion does not apply to patients with bilateral ovarian resection and/or hysterectomy or postmenopausal patients).

-

Exclusion Criteria:

Subjects who have received radiotherapy, chemotherapy, immunosuppressive agents, monoclonal antibodies, oral epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs), or anti-angiogenic drugs within the past six months.

Subjects who have participated in another interventional clinical trial, undergone major surgical procedures, or scheduled for surgery within 30 days prior to screening.

Patients with severe underlying diseases that preclude tolerance to the treatment.

History of other malignancies, except for cured cervical carcinoma in situ, skin basal cell carcinoma, or malignancies cured for more than 5 years without recurrence.

Presence of uncontrolled comorbidities such as heart failure, diabetes mellitus, hypertension, thyroid disorders, psychiatric illnesses, etc.

Subjects with contraindications to immunotherapy, including those with immune dysfunction diseases (such as rheumatoid arthritis, psoriasis, systemic lupus erythematosus, HIV infection, hepatitis B, hepatitis C, chronic use of steroids for autoimmune diseases), recipients of allogeneic transplants, patients with interstitial lung disease, or those with meningeal metastasis or progressive brain metastasis.

Allergy to any of the drugs or their components used in the study protocol. Grade 2 or higher peripheral neuropathy or hearing loss according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

Pregnant women (confirmed by blood or urine human chorionic gonadotropin [HCG] test) or lactating mothers, or subjects of reproductive age who are unwilling or unable to adopt effective contraceptive measures until at least 6 months after the last treatment in the study.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
ORR[RECIST1.1] | 3 months
  objective response rate assessed by RECIST 1.1

SECONDARY OUTCOMES:
mPFS | 1 year
  median progression-free survival assessed by RECIST 1.1
OS | 2 years
  median overall survival
2-year PFS rate | 2 years
  2-year progression-free survival rate assessed by RECIST 1.1
DCR | 3 months
  disease control rate assessed by RECIST 1.1
DOR | 2 years
  duration of response assessed by RECIST 1.1
adverse event | 3 years
  incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: He Xiaohui, Principal Investigator — Department of Medical Oncology
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medcial Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No